CLINICAL TRIAL: NCT05493852
Title: A Real-world Study of the FARAPULSE Pulsed Field Ablation System in A Chinese Population With Paroxysmal Atrial Fibrillation
Brief Title: A RWS of the FARAPULSE in A Chinese Population With PAF
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PF109
Record Dates: First submitted 2022-08-02; First posted 2022-08-09 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FARAPULSE Pulsed Field Ablation System: Patients diagnosed as paroxysmal atrial fibrillation with indication of ablation.
  Interventions: Device: FARAPULSE Pulsed Field Ablation System

INTERVENTIONS:
Device: FARAPULSE Pulsed Field Ablation System — Patients diagnosed as paroxysmal atrial fibrillation with indication of ablation will be treated by FARAPULSE Pulsed Field Ablation System.

SUMMARY:
The real world study is a retrospective and/or prospective, single-center, single-arm observational study to observe the safety and effectiveness of the FARAPULSE Pulsed Field Ablation System for treatment of recurrent, symptomatic Paroxysmal Atrial Fibrillation (PAF) in a Chinese population.

DETAILED DESCRIPTION:
The primary effectiveness endpoint is the acute procedural success, defined as the proportion of subjects that achieve electrical isolation of all PVs using FARAPULSE Pulsed Field Ablation system only.

The primary safety endpoint is defined as the occurrence of the acute serious procedure-related and /or device-related adverse events at 7 days post index procedure.

Primary endpoints analysis is planned to be conducted after all enrolled subjects have completed data collection at 1-month follow-up visit. All the subjects underwent study device treatment will be followed up to 12 months after the procedure, and the secondary and other endpoints will be analyzed then.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are ≥ 18 and ≤ 75 years of age on the day of enrollment;
2. Subjects whose preoperative diagnosis is PAF confirmed by the clinician;
3. De novo ablation procedure for PAF with Class I or IIa recommendations* according to 2018 Chinese expert consensus on atrial fibrillation therapy;
4. Subjects who are able and willing to provide the defined observational data and/or participate in baseline and follow-up evaluations for the full study;
5. Subjects who are willing and capable of providing informed consent.

Exclusion Criteria:

1. Subjects who, in the judgment of the investigator, have a life expectancy of less than one year before the procedure;
2. Women of childbearing potential who are, or plan to become, pregnant during the time of the study;
3. Subjects with any known contraindication to AF ablation with FARAPULSE Pulsed Field Ablation system, anticoagulation therapy, or contrast media in the judgment of the investigator or subjects unwillingness to use systemic anticoagulation
4. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as paroxysmal atrial fibrillation with indication of ablation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minglong Chen, Dr, Principal Investigator — Boao Super Hospital
Locations (1):
- Boao Super Hospital, Bo'ao, Hainan, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FARAPULSE Pulsed Field Ablation System
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FARAPULSE Pulsed Field Ablation System
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 57.6 [32 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 30
Height [Mean (Full Range); unit: cm] | 165.4 [145 to 183]
BMI [Mean (Full Range); unit: kg/m^2] | 25.3 [16.5 to 30.2]
Weight [Mean (Full Range); unit: Kg] | 70 [34.6 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Procedural Success
Description: The primary effectiveness endpoint is the acute procedural success, defined as the proportion of subjects that achieve electrical isolation of all PVs using FARAPULSE Pulsed Field Ablation system only.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Pulsed Field Ablation System
Number analyzed (Participants) | 30
Participants | 30

2. Primary Outcome: Number of Participants With SAE Related to the Procedure or Device at 7 Days Post Index Procedure
Description: The primary safety endpoint is defined as the occurrence of the acute serious procedure-related and /or device-related adverse events at 7 days post index procedure.
Time Frame: 7 Days
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Pulsed Field Ablation System
Number analyzed (Participants) | 30
Participants | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | FARAPULSE Pulsed Field Ablation System
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 20/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Pulsed Field Ablation System (N=30)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Pulsed Field Ablation System (N=30)
Myocardial injury (Cardiac disorders) | 5 (5)
Supraventricular extrasystoles (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Puncture site haematoma (General disorders) | 2 (2)
Catheter site haematoma (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Puncture site pain (General disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Blood glucose increased (Investigations) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT05493852/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT05493852/SAP_001.pdf